CLINICAL TRIAL: NCT04478682
Title: The Effect of Continuous Breastfeeding Support Provided to Mothers Through WhatsApp Messaging Application on Breastfeeding: A Randomized Controlled Trial
Brief Title: Breastfeeding Support Provided to Mothers Through WhatsApp Messaging Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Sevda KORKUT ÖKSÜZ, Research Assistant, Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AhiEvranU
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Exclusive Breastfeeding; Breastfeeding Support
Keywords: Breastfeeding support; Exclusive breastfeeding; WhatsApp messaging application; Motivation; Attitude
MeSH Terms: conditions — Breast Feeding; Behavior

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WhatsApp Messaging Application (Experimental): Continuous breastfeeding support will be provided for the first 6 months through WhatsApp messaging application. Mothers will be contacted once a week through WhatsApp and feedback will be received on the breastfeeding process. The questions of the mother regarding breastfeeding will be answered by text / voice message or video call.
  Interventions: Other: Breastfeeding Support Provided to Mothers Through WhatsApp Messaging Application
- Standard breastfeeding support (No Intervention): She will receive standard breastfeeding support after delivery. Breastfeeding will not receive continuous breastfeeding support for the first 6 months after discharge.

INTERVENTIONS:
Other: Breastfeeding Support Provided to Mothers Through WhatsApp Messaging Application — Breastfeeding support provided to mothers through WhatsApp messaging application will be maintained for the first 6 months after birth. In the first 1 month, standard information sharing will be made through whatsApp. Also, for the first 6 months, solutions generating shares will be made according to the problems and questions of the mother regarding breastfeeding.
  Arms: WhatsApp Messaging Application

SUMMARY:
The research was planned as a randomized controlled experimental study in order to determine the effect of continuous breastfeeding support provided to mothers through WhatsApp messaging application on breastfeeding.

Research Hypotheses H0: Continuous breastfeeding support provided to mothers through WhatsApp messaging application has no effect on breastfeeding.

H1: Continuous breastfeeding support provided to mothers through WhatsApp messaging application increases the rate of exclusive breastfeeding.

H2: Continuous breastfeeding support provided to mothers through WhatsApp messaging application increases the breastfeeding duration of the mothers.

H3: Continuous breastfeeding support provided to mothers through WhatsApp messaging application reduces the rate of mothers giving their babies other foods than breast milk.

H4: Continuous breastfeeding support provided to mothers through WhatsApp messaging application reduces bottle feeding rates.

H5: Continuous breastfeeding support provided to mothers through WhatsApp messaging application reduces the rate of pacifier use.

H6: Continuous breastfeeding support provided to mothers through WhatsApp messaging application reduces the incidence of mothers' breastfeeding problems.

H7: Continuous breastfeeding support provided to mothers through WhatsApp messaging application affects mothers' breastfeeding attitude positively.

H8: Continuous breastfeeding support provided to mothers through WhatsApp messaging application increases the motivation of breastfeeding mothers.

DETAILED DESCRIPTION:
METHOD:

Place of the Research:

The data of the research will be collected in the postpartum service of Zeynep Kamil Women And Chıldren Dıseases Tranıng And Research Hospıtal in Istanbul. After then 6 months of follow-up will be continued trough WhatsApp application.

The Universe and the Sample of the Research:

The universe of the research; It will comprise primipa mothers and babies who are hospitalized in the postpartum ward of the specified dates, deliver vaginal or cesarean delivery, and meet the sample selection criteria.

The sample of the research was determined by statistic analysis by power analysis. Power analysis was performed by using G * Power (v3.1.7) program to determine the number of samples. The power of the study is expressed as 1-β (olasılığı = type II error probability) and research should generally have 80% power. According to Cohen's effect size coefficients; Assuming that the evaluations to be made between the two independent groups will have a medium effect size (d = 0.5), considering the fact that there should be at least 64 people in the groups and there may be losses in the working process, each group decided to recruit 70 people. 140 people in total. it is given. Computerized randomization method will be used in the research.

In the collection of research data; Mother and Newborn Data Collection Form Postpartum Breastfeeding Evaluation and Follow-up Form Application Satisfaction Evaluation Form Breastfeeding Attitudes of The Evaluation Scale Primipara Breastfeeding Motivation Scale (PBMS) 5 data collection forms will be used.

Application of the research:

The researcher will briefly talk about the scope and content of the research by meeting with the mothers who meet the case selection criteria. Written consents will be obtained through the "Informed Volunteer Consent Form" asking mothers whether they want to participate in the study. Mothers who wish to participate in the study will be randomly determined by computer-assisted randomization method. Applications made after randomization will be carried out with the following steps; Experimental group; Information will be obtained from the mothers who agreed to participate in the study in line with the "Mother and Newborn Data Total Form", Mothers participating in the study will receive routine breastfeeding training at the hospital after birth, The breastfeeding attitude of the mother will be evaluated with the "Breastfeeding Attitude Scale", and the breastfeeding motivation of the mother will be evaluated with the "Breastfeeding Motivation Scale", In line with the needs of the mothers, breastfeeding support and motivation will be provided, In the first 1 month, basic standard information sharing (see "Basic Standard Information Sharing") will be made determined by the researcher. Later, information sharing will be made regarding the questions and problems of the mother, Individual breastfeeding support provided to mothers through WhatsApp will continue for 6 months, Mothers will be contacted once a week through WhatsApp and feedback will be received on the breastfeeding process, The questions of the mother regarding breastfeeding will be answered by text / voice message or video call, In the postpartum period (day 7, day 15, month 1, month 2, month 4 and month 6) mothers will be called by phone. Breastfeeding conditions will be evaluated with "Postpartum Breastfeeding Evaluation and Follow-up Form".

Breastfeeding attitudes of the mothers will be assessed with the Breastfeeding Attitudes of the Evaluation Scale" before breastfeeding education in hospital and through online survey at the 6th Month.

Breastfeeding motivations of the mothers will be assessed with the " Primipara Breastfeeding Motivation Scale " through online survey at the 6th Month.

The mothers' satisfaction with the continuous breastfeeding support provided through WhatsApp will be evaluated with the "Application Satisfaction Evaluation Form" through online survey.

Basic Standard Information Sharing; New coronavirus (COVID-19) and breastfeeding Suggestion on breastfeeding (motivational-enhancing videos that emphasize breastfeeding is instinctive) The importance of breast milk (positive effects on mother and baby will be explained) Sharing of health institutions emphasizing the importance of breastfeeding (WHO, UNICEF, Ministry of Health) Milk production of breasts (Frequent breastfeeding will be supported by videos) Baby holding the breast (Mothers will be emphasized that the baby's sucking ability instinctively and will be supported with videos) Skin-to-skin contact and breastfeeding Reasons for breastfeeding only for the first 6 months Symptoms that show that the baby is sucking effectively Control Group; Information will be obtained from the mothers who agreed to participate in the study in line with the "Mother and Newborn Data Total Form", Mothers participating in the study will receive routine breastfeeding training at the hospital after birth, The breastfeeding attitude of the mother will be evaluated with the "Breastfeeding Attitude Scale", and the breastfeeding motivation of the mother will be evaluated with the "Breastfeeding Motivation Scale", In line with the needs of the mothers, breastfeeding support and motivation will be provided, In the postpartum period (day 7, day 15, month 1, month 2, month 4 and month 6) mothers will be called by phone. Breastfeeding conditions will be evaluated with "Postpartum Breastfeeding Evaluation and Follow-up Form".

Breastfeeding attitudes of the mothers will be assessed with the Breastfeeding Attitudes of the Evaluation Scale" before breastfeeding education in hospital and through online survey at the 6th Month.

Breastfeeding motivations of the mothers will be assessed with the " Primipara Breastfeeding Motivation Scale " through online survey at the 6th Month.

Analysis:

NCSS (Number Cruncher Statistical System) 2007 (Kaysville, Utah, USA) program will be used for statistical analysis of the research. Statistical significance will be accepted as p <0.05.

ELIGIBILITY:
Inclusion Criteria:

For the mother;

* 18 years and older
* Primipar,
* Having healthy pregnancy and uncomplicated birth,
* No health problems preventing breastfeeding (drug use, HIV, etc.),
* Not having any obstacle to communication (not knowing Turkish, mental retardation etc.),
* Being literate,
* Having a smart phone and internet connection,
* It was determined to be able to use WhatsApp application. For baby;
* Being healthy and term
* No health problems preventing breastfeeding (Esophageal atresia, cleft palate, cleft lip etc.)
* Its weight is between 2500-4000 gr.
* It was determined that the Apgar Score was above 7.

Exclusion Criteria:

* Mothers with multiple pregnancies,
* Infants lying in NICU due to health problems in the postpartum period will be excluded from the scope of the research.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 18 years and older who primiparous women who gave birth
Enrollment: 150 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Attitudes of The Evaluation Scale | In our study, will be applied before breastfeeding education in hospital and through online survey at postpartum 6th months for both groups
  This scale assesses various aspects of attitudes that direct mothers' breastfeeding behavior. Examines breastfeeding as behavior.
  The scale is a five-point Likert type consisting of 46 items, easy to apply, and which people can answer on their own, and it can be applied to all mothers. Some items in the scale (3, 4, 6, 7, 8, 11, 13, 15, 19, 23, 24, 26, 27, 28, 29, 30, 31, 32, 37, 38, 42, 43) As a positive attitude, I agree with the statement "I totally disagree" to 4-3-2-1-0, while some items (1, 2, 5, 9, 10, 12, 14, 16, 17, 18, 20, 21 (22, 25, 33, 34, 35, 36, 39, 40, 41, 44, 45, 46) are considered negative, and the opposite score is scored as 0-1-2-3-4 from the statement entirely agree. In this way, the total score that can be obtained from the scale is between 0 and 184. As the score increases, breastfeeding attitude is evaluated as positive.
Primipara Breastfeeding Motivation Scale (PBMS) | at postpartum 6th months through online survey for both groups
  This scale evaluates postpartum breastfeeding motivation level in primiparous. The scale consists of 24 items in total. After applying to the sample group, the factor analysis of the scale was made and it was determined to have 5 factors.
  1. Intrinsic motivation and integrated regulation
  2. Identified regulation
  3. Mirrored editing
     External regulation is examined in two sub-dimensions:
  4. External regulation (instrumental needs)
  5. External regulation (baby health) Scale items are rated from 1 = Never disagree to 4 = Strongly agree. The scale is in 4-point Likert type, and each item is scored between 1-4. The scale does not have a total score. The score of the sub-dimensions is calculated by taking the average of the scale sub-dimension scores. As the score obtained from the sub-dimension of the scale increases, the motivation representing that sub-dimension increases.
Application Satisfaction Evaluation Form | at postpartum 6th months through online survey for only experimental group
  Evaluates the satisfaction of mothers from breastfeeding support provided through WhatsApp messaging application.
  It is a form consisting of 10 questions by the researcher to evaluate the satisfaction of the mothers from the breastfeeding support given through the social media group (WhatsApp) by making use of the literature information.
  The answer to each question will be evaluated as yes / no. In the tenth question, he will be asked to score the application. There will be a minimum of 1 and a maximum of 10 points.

CONTACTS AND LOCATIONS:
Overall Officials: Sevda KORKUT ÖKSÜZ, R.A, Principal Investigator — Kirsehir Ahi Evran Universitesi
Locations (1):
- Zeynep Kamil Women And Chıldren Dıseases Tranıng And Research Hospıtal, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balaguer Martinez JV, Valcarce Perez I, Esquivel Ojeda JN, Hernandez Gil A, Martin Jimenez MDP, Bernad Albareda M. [Telephone support for breastfeeding by primary care: a randomised multicentre trial]. An Pediatr (Engl Ed). 2018 Dec;89(6):344-351. doi: 10.1016/j.anpedi.2018.02.007. Epub 2018 Mar 22. Spanish. PMID 29576447
- [Background] Reiss K, Andersen K, Barnard S, Ngo TD, Biswas K, Smith C, Carpenter J, Church K, Nuremowla S, Pearson E. Using automated voice messages linked to telephone counselling to increase post-menstrual regulation contraceptive uptake and continuation in Bangladesh: study protocol for a randomised controlled trial. BMC Public Health. 2017 Oct 3;17(1):769. doi: 10.1186/s12889-017-4703-z. PMID 28974209
- [Background] Simonetti V, Palma E, Giglio A, Mohn A, Cicolini G. A structured telephonic counselling to promote the exclusive breastfeeding of healthy babies aged zero to six months: a pilot study. Int J Nurs Pract. 2012 Jun;18(3):289-94. doi: 10.1111/j.1440-172X.2012.02040.x. PMID 22621300
- [Background] Cavalcanti DS, Cabral CS, de Toledo Vianna RP, Osorio MM. Online participatory intervention to promote and support exclusive breastfeeding: Randomized clinical trial. Matern Child Nutr. 2019 Jul;15(3):e12806. doi: 10.1111/mcn.12806. Epub 2019 Apr 11. PMID 30825414
- [Background] Kapinos K, Kotzias V, Bogen D, Ray K, Demirci J, Rigas MA, Uscher-Pines L. The Use of and Experiences With Telelactation Among Rural Breastfeeding Mothers: Secondary Analysis of a Randomized Controlled Trial. J Med Internet Res. 2019 Sep 3;21(9):e13967. doi: 10.2196/13967. PMID 31482848
- [Background] Durmaz S, Ergin I, Durusoy R, Hassoy H, Caliskan A, Okyay P. WhatsApp embedded in routine service delivery for smoking cessation: effects on abstinence rates in a randomized controlled study. BMC Public Health. 2019 Apr 8;19(1):387. doi: 10.1186/s12889-019-6727-z. PMID 30961557
- [Derived] Sevda KO, Sevil I. Continuous Lactation Support Provided Through the WhatsApp Messaging Application: A Randomized Controlled Trial. J Hum Lact. 2023 Nov;39(4):666-678. doi: 10.1177/08903344231192948. Epub 2023 Aug 30. PMID 37646262